CLINICAL TRIAL: NCT02963233
Title: Type II Pediatric Supracondylar Humerus Fracture Management and Outcomes: A Prospective Multi-centre Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Children's Hospital (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Principal Investigator, Christopher Reilly, Associate Professor, University of British Columbia
Other Study IDs: H15-00835
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Trauma; Fracture;Elbow
MeSH Terms: conditions — Wounds and Injuries; Elbow Fractures | interventions — Immobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-operative Group: Patients treated within the non-operative group will be treated with gentle reduction by the orthopaedic surgery team in the emergency department under procedural sedation. Immobilization and maintenance of reduction will be obtained through either taping of the elbow in a flexed (100-110 degree) and pronated position or through long-arm casting at 90 degrees of flexion. Immobilization type and position will be noted.
  Interventions: Procedure: Non-operative reduction and immobilization
- Operative Group: Patients treated operatively will be largely treated with closed reduction and percutaneous pinning with 2-3 laterally-based k-wires, followed by long-arm immobilization. Immobilization type and position will be noted.
  Interventions: Procedure: Closed reduction and percutaneous pinning and immobilization

INTERVENTIONS:
Procedure: Closed reduction and percutaneous pinning and immobilization
  Groups: Operative Group
Procedure: Non-operative reduction and immobilization
  Groups: Non-operative Group

SUMMARY:
The treatment of pediatric supracondylar humerus fractures is controversial, but despite the injury's high incidence there is a lack of high level evidence to guide operative versus non-operative decision making for displaced fractures with an intact posterior cortex (Gartland Type II). This study aims to prospectively compare clinical, functional, and radiographic outcomes between operatively and non-operatively treated patients using a prospective multi-centre cohort design.

DETAILED DESCRIPTION:
Purpose:

The purpose of this prospective multi-center observational study is to compare the clinical, functional, and radiographic parameters and outcomes between operatively and non-operatively treated Type II supracondylar humerus fractures in skeletally immature patients. The secondary aim of the study is to develop and deploy an effective pediatric orthopaedic elbow trauma database as part of the Canadian Pediatric Orthopaedic Group (CPOG) that can be used to prospectively collect multi-center anonymized patient data and functional outcomes.

Hypothesis:

We hypothesize that non-operative treatment will be non-inferior to operative treatment.

Justification:

The extension-type pediatric supracondylar humerus fracture is the most common fracture about the elbow in the skeletally immature population and among the most common fractures requiring operative intervention in children (Carson 2006, Abzug 2012). Despite being the subject of extensive study, there are few prospective studies and none that look specifically at the Gartland Type II extension-type fracture and that compare operative and non-operative treatment protocols (AAOS CPG 2011). The current evidence for the treatment of these fracture sub-types is low, but clinical opinions regarding treatment method are strong. This has led to a clinical practice vs. evidence mismatch.

The existing level of evidence does not support the strong clinical opinions on the treatment of this fracture pattern, and given its significant prevalence this is an area that requires objective prospective study. A finding of a significant clinical effect difference would guide future treatment of this common entity, while a finding of clinical equipoise could allow for the development of a well designed and focused prospective randomized controlled trial.

Research Methods:

The study is designed as a multi-center, observational, cohort protocol with an initial focus on the comparison of outcomes between several Canadian pediatric academic centers with contrasting (operative and non-operative) general approaches to the management of isolated closed extension-type Gartland Type II supracondylar humerus fractures.

Patients treated within the non-operative group will be treated with gentle reduction by the orthopaedic surgery team in the emergency department under procedural sedation. Immobilization and maintenance of reduction will be obtained through either taping of the elbow in a flexed (100-110 degree) and pronated position or through long-arm casting at 90 degrees of flexion. Immobilization type and position will be noted. Patients treated surgically will be largely treated with closed reduction and percutaneous pinning with 2-3 laterally-based k-wires, followed by long-arm immobilization. Continued care and follow-up practices will be the same across treatment groups, as outlined below under "Study Visits".

The null hypothesis is that non-operative treatment of Type II supracondylar humerus fractures is inferior to closed reduction and percutaneous pinning.

Evaluation of Outcomes and Variables:

Demographics such as age, sex, handedness, and mechanism of injury will be recorded. Radiographic parameters measured will include stratification into Type IIA vs IIB fractures, and angular deformity and displacement through the lateral humeral capitellar angle (LHCA) and Baumann's angle. These will be captured at each clinical visit, including pre- and post-reduction. On the lateral radiograph, the LHCA is measured as the angle between the anterior humeral line and a line perpendicular to the capitellar physis (ie. a line through the long axis of the capitellar ossific nucleus). A lateral humeral capitellar angle less than 20 degrees or a change of greater than 10 degrees over time will be considered significant. A Baumann's angle outside the accepted norm of 9-26 degrees, or a change over time of greater than 6 degrees will be considered significant. In addition, the pre-reduction and post-reduction Gordon index (a radiographic measure of lateral rotation through the fracture site on the lateral radiograph) will be measured, as will the Griffet index which expands upon the same concept using also the AP radiograph (Griffet 2004). De-identified radiographs will also be uploaded where techinically feasible to the central database, where radiographic parameters can be re-assessed by a blinded third party. Clinical outcomes will be judged based on healing, return to activities, and range of motion. Any complications encountered will be recorded. Functional outcomes will be judged via the Flynn criteria for both functional and cosmetic outcome (Flynn 1974, Cheng 1995). The PODCI upper extremity score (Daltroy 1998) and the QuickDASH (Kennedy 2011) will also be used.

Primary Outcome: Change in Lateral Humerocapitellar Angle (LHCA) Change in the LHCA over the period of immobilization is the primary outcome being measured in this study, and will be measured on all radiographs. Maintenance of fracture reduction is assessed by the change in the LHCA between these two radiographs. This angle primarily assesses the reduction in the sagittal plane and thus is most sensitive to flexion and extension. The normal LHCA is considered to be 30 degrees of anterior angulation. It has been shown that with changes of less than 10 degrees, good elbow function can still be expected. Using a single measurement of the LHCA at the completion of treatment would fail to account for the quality of the initial reduction but using a change in the LHCA controls for this additional variability. Also, using clinical measures would require waiting until maximum range of motion of the elbow is regained and this would introduce the variability associated with remodeling and rehabilitation and would not accurately reflect the efficacy of the immobilization method itself. Although a standardized method for obtaining the lateral radiograph will be employed in all study patients, it has been noted that the LHCA can vary significantly if there is humeral rotation on the radiograph. For this reason, the quality of the radiograph will also be recorded after assessing the superimposition of the posterior supracondylar ridges. Perfect superimposition of the supracondylar ridges indicates a true lateral of the distal humerus.

Secondary Endpoints: Baumann's Angle, Flynn's Elbow Score, Conversion to Operative treatment, Revision Operation, Complications Baumann's angle is that formed between the physeal line of the lateral condyle and a line perpendicular to the long axis of the humerus as seen on anteroposterior radiographs of the elbow. Change in the angle over time will be measured. This angle can be used to detect varus angulation of the distal part of the humerus. A normal angle is in the range of 9° to 26°. The Baumann angle has been shown to vary 6° for every 10° of humeral rotation on the anteroposterior radiograph. Thus a difference of 6° between the post-reduction and final Baumann angles has been empirically chosen to represent a meaningful change. This allows for minor variations in arm positioning during the radiographic evaluation as well as measurement variability.

Flynn's elbow score accounts for both elbow function and cosmesis. Elbow function is measured in degrees of lost flexion and/or extension compared to the opposite elbow. Elbow cosmesis is measured by the change in carrying angle compared to the opposite elbow. These are rated as excellent (0-5°), good (6-10°), fair (11-15°) and poor (>15°). Overall results are determined by the worst grade in functional and cosmetic ratings.

Patients requiring operative intervention after failing non-operative treatment, as well as those requiring revision operation, will have such results and their clinical contexts recorded. Complications, both objectively observed by the clinical team as well as those subjectively experienced by patients and families will likewise be assessed and recorded.

Statistical Analysis:

It is estimated based on a power analysis and sample size calculation assessing for non-inferiority of non-operative management that a minimum total of 36 (18 patients in each cohort) patients will be needed for this study. This sample size is based on a one-tailed t-test for independent means, with α=0.05, β=0.1 (power of 0.90). A significant difference is considered to be within 6 degrees of change in the LHCA (Lateral Humeral Capitellar Angle) between the operative and non-operative groups, as differences of 5 degrees or less on elbow radiographs are considered to be within measurement error. The measurement error is expected to be the same in both groups. Estimations of means and standard deviations of LHCA were based on recent local research (Roberts 2014) . Using an online institutional power and sample size calculator (Brant 2014) which is based on standard two-sample inference estimation of sample size and power for comparing two means, the investigators developed a table with various iterations of possible calculations. Erring on the conservative, the investigators have chosen to accept a sample size of 18 patients in each group.

Baseline demographics and characteristics will be summarized using standard summary statistics. Continuous variables will be expressed in terms of means and standard deviations, and categorical variables will be summarized in terms of frequency and percentages. A one-sided student's t-test will be used for comparison between primary outcomes of the study cohorts, for non-inferiority. All statistical tests will be performed at an α-level of 0.05. Multi-variate regression analyses will be performed to assess for other variables affecting outcomes. Sub-group analyses will be undertaken to assess for within group differences.

Based on our power analysis and sample size calculations, and a conservative projected drop out rate of 20%, the investigators conclude that a minimum of 23 patients per treatment group (18 subjects divided by 0.8 to account for projected drop out) need to be recruited to effectively prove non-inferiority. That said, given that the investigators plan to also pursue as secondary measures multi-variate analyses and sub-group analyses, the plan is to improve our likelihood of obtaining significance by aiming for a minimum recruitment of 30 patients per cohort, for a total minimum number of patients of 60.

By using a multi-centre methodology, the investigators hope to be able to not only meet but also significantly exceed our minimum recruitment requirements. This should serve the dual purpose of adding variability in care environments and providers and therefore improve generalizability of results, as well as strengthen our statistical significance particularly with our secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-12 years
* Isolated supracondylar humerus fracture
* Gartland Type II extension-type fracture
* Closed injury

Exclusion Criteria:

* Neurovascular compromise
* Underlying musculoskeletal disorder

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients identified with a closed, isolated Gartland Type II extension-type supracondylar humerus fracture between 2-12 years, recruited within their acute treatment phase between initial injury presentation either to the emergency department or the orthopaedic clinic and 6 weeks post-injury.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in Lateral Humerocapitellar Angle | 3 months
  Change in the LHCA over the period of immobilization is the primary outcome being measured in this study, and will be measured on all radiographs. Maintenance of fracture reduction is assessed by the change in the LHCA between these two radiographs. This angle primarily assesses the reduction in the sagittal plane and thus is most sensitive to flexion and extension. The normal LHCA is considered to be 30 degrees of anterior angulation. It has been shown that with changes of less than 10 degrees, good elbow function can still be expected.

SECONDARY OUTCOMES:
Baumann's Angle | 3 months
  Baumann's angle is that formed between the physeal line of the lateral condyle and a line perpendicular to the long axis of the humerus as seen on anteroposterior radiographs of the elbow. Change in the angle over time will be measured. This angle can be used to detect varus angulation of the distal part of the humerus. A normal angle is in the range of 9° to 26°. The Baumann's angle has been shown to vary 6° for every 10° of humeral rotation on the anteroposterior radiograph. Thus a difference of 6° between the post-reduction and final Baumann angles has been empirically chosen to represent a meaningful change. This allows for minor variations in arm positioning during the radiographic evaluation as well as measurement variability.
Flynn's Elbow Score | 1 year
  Flynn's elbow score accounts for both elbow function and cosmesis. Elbow function is measured in degrees of lost flexion and/or extension compared to the opposite elbow. Elbow cosmesis is measured by the change in carrying angle compared to the opposite elbow. These are rated as excellent (0-5°), good (6-10°), fair (11-15°) and poor (>15°). Overall results are determined by the worst grade in functional and cosmetic ratings.

OTHER OUTCOMES:
Complications/Conversion to Operative Treatment/Revision Operation | 1 year
  Patients requiring operative intervention after failing non-operative treatment, as well as those requiring revision operation, will have such results and their clinical contexts recorded. Complications, both objectively observed by the clinical team as well as those subjectively experienced by patients and families will likewise be assessed and recorded.

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (13):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Prince George Surgery Centre, Prince George, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Janeway Children's Hospital, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - La Cité Médical Québec, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulpuri K, Hosalkar H, Howard A. AAOS clinical practice guideline: the treatment of pediatric supracondylar humerus fractures. J Am Acad Orthop Surg. 2012 May;20(5):328-30. doi: 10.5435/JAAOS-20-05-328. No abstract available. PMID 22553105
- [Background] Abzug JM, Herman MJ. Management of supracondylar humerus fractures in children: current concepts. J Am Acad Orthop Surg. 2012 Feb;20(2):69-77. doi: 10.5435/JAAOS-20-02-069. PMID 22302444
- [Background] Bashyal RK, Chu JY, Schoenecker PL, Dobbs MB, Luhmann SJ, Gordon JE. Complications after pinning of supracondylar distal humerus fractures. J Pediatr Orthop. 2009 Oct-Nov;29(7):704-8. doi: 10.1097/BPO.0b013e3181b768ac. PMID 20104149
- [Background] Blasier RD. Gartland type-II supracondylar humeral fractures in children: commentary on an article by Luis Moraleda, MD, et al.: "Natural history of unreduced Gartland type-II supracondylar fractures of the humerus in children. a two to thirteen-year follow-up study". J Bone Joint Surg Am. 2013 Jan 2;95(1):e7. doi: 10.2106/jbjs.l.01324. No abstract available. PMID 23405412
- [Background] Carson S, Woolridge DP, Colletti J, Kilgore K. Pediatric upper extremity injuries. Pediatr Clin North Am. 2006 Feb;53(1):41-67, v. doi: 10.1016/j.pcl.2005.10.003. PMID 16487784
- [Background] Cheng JC, Lam TP, Shen WY. Closed reduction and percutaneous pinning for type III displaced supracondylar fractures of the humerus in children. J Orthop Trauma. 1995;9(6):511-5. doi: 10.1097/00005131-199509060-00009. PMID 8592265
- [Background] Daltroy LH, Liang MH, Fossel AH, Goldberg MJ. The POSNA pediatric musculoskeletal functional health questionnaire: report on reliability, validity, and sensitivity to change. Pediatric Outcomes Instrument Development Group. Pediatric Orthopaedic Society of North America. J Pediatr Orthop. 1998 Sep-Oct;18(5):561-71. doi: 10.1097/00004694-199809000-00001. PMID 9746401
- [Background] Fitzgibbons PG, Bruce B, Got C, Reinert S, Solga P, Katarincic J, Eberson C. Predictors of failure of nonoperative treatment for type-2 supracondylar humerus fractures. J Pediatr Orthop. 2011 Jun;31(4):372-6. doi: 10.1097/BPO.0b013e31821adca9. PMID 21572273
- [Background] Flynn JC, Matthews JG, Benoit RL. Blind pinning of displaced supracondylar fractures of the humerus in children. Sixteen years' experience with long-term follow-up. J Bone Joint Surg Am. 1974 Mar;56(2):263-72. No abstract available. PMID 4375679
- [Background] Hadlow AT, Devane P, Nicol RO. A selective treatment approach to supracondylar fracture of the humerus in children. J Pediatr Orthop. 1996 Jan-Feb;16(1):104-6. doi: 10.1097/00004694-199601000-00021. PMID 8747365
- [Background] Lins RE, Simovitch RW, Waters PM. Pediatric elbow trauma. Orthop Clin North Am. 1999 Jan;30(1):119-32. doi: 10.1016/s0030-5898(05)70066-3. PMID 9882730
- [Background] Moraleda L, Valencia M, Barco R, Gonzalez-Moran G. Natural history of unreduced Gartland type-II supracondylar fractures of the humerus in children: a two to thirteen-year follow-up study. J Bone Joint Surg Am. 2013 Jan 2;95(1):28-34. doi: 10.2106/jbjs.l.00132. PMID 23405411
- [Background] Omid R, Choi PD, Skaggs DL. Supracondylar humeral fractures in children. J Bone Joint Surg Am. 2008 May;90(5):1121-32. doi: 10.2106/JBJS.G.01354. PMID 18451407
- [Background] O'Hara LJ, Barlow JW, Clarke NM. Displaced supracondylar fractures of the humerus in children. Audit changes practice. J Bone Joint Surg Br. 2000 Mar;82(2):204-10. PMID 10755427
- [Background] Parikh SN, Wall EJ, Foad S, Wiersema B, Nolte B. Displaced type II extension supracondylar humerus fractures: do they all need pinning? J Pediatr Orthop. 2004 Jul-Aug;24(4):380-4. doi: 10.1097/00004694-200407000-00007. PMID 15205619
- [Background] Pirone AM, Graham HK, Krajbich JI. Management of displaced extension-type supracondylar fractures of the humerus in children. J Bone Joint Surg Am. 1988 Jun;70(5):641-50. PMID 3392056
- [Background] Roberts L, Strelzow J, Schaeffer EK, Reilly CW, Mulpuri K. Nonoperative Treatment of Type IIA Supracondylar Humerus Fractures: Comparing 2 Modalities. J Pediatr Orthop. 2018 Nov/Dec;38(10):521-526. doi: 10.1097/BPO.0000000000000863. PMID 27636909
- [Background] Williamson DM, Cole WG. Treatment of selected extension supracondylar fractures of the humerus by manipulation and strapping in flexion. Injury. 1993 Apr;24(4):249-52. doi: 10.1016/0020-1383(93)90180-e. PMID 8325683
- See also: Brant R. Inference for Means: Comparing Two Independent Samples. University of British Columbia, Department of Statistics. http://www.stat.ubc.ca/~rollin/stats/ssize/n2.html Last accessed Oct 31, 2014. — http://www.stat.ubc.ca/~rollin/stats/ssize/n2.html